CLINICAL TRIAL: NCT07311434
Title: Evaluation of Perceived Outcomes With AGZ: A Randomized, Controlled, Consumer Perception Study
Brief Title: Sleep and Morning Wellbeing Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Athletic Greens International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AGZ001
Record Dates: First submitted 2025-12-18; First posted 2025-12-31 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Sleep; Relaxation; Stress; Daytime Sleepiness
MeSH Terms: conditions — Disorders of Excessive Somnolence

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Supplement (Experimental): Sleep Supplement
  Interventions: Dietary Supplement: Sleep Supplement
- Usual Diet (No Intervention): Usual Diet

INTERVENTIONS:
Dietary Supplement: Sleep Supplement — Powdered sleep supplement
  Arms: Sleep Supplement

SUMMARY:
The study will be a prospective randomized, controlled clinical study. There will be interventional treatment for a total of 30 days. The subjects will complete questionnaires throughout the study at pre-specified timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age 25-59 years.
* BMI ≥18.5 and ≤29.9 kg/m².
* Currently experiencing issues with sleep quality, falling asleep, staying asleep, or waking during the night.
* RU-SATED score ≤17.
* Willing and able to follow the study protocol.
* Willing to discontinue any other supplements (including nootropics, adaptogens, calming herbs), medications, herbal remedies, or over-the-counter sleep medications (e.g., zolpidem, diphenhydramine, Benadryl, ZzzQuil, Unisom, magnesium or melatonin products) used to assist with sleep during the study.
* Agree to limit alcohol intake within approximately 4 hours of bedtime throughout participation.
* Agree to limit caffeine intake to ≤400 mg/day (about 3-4 cups of coffee) and avoid ingestion of caffeine-containing products after 2:00 PM during the study period.
* Generally healthy and not living with any uncontrolled chronic disease.
* Resides in the United States.
* Willing to discontinue any restricted products and adhere to all required study assessments.

Exclusion Criteria:

* Diagnosed chronic sleep conditions (e.g., insomnia, narcolepsy, REM Behavior Disorder, moderate to severe restless leg syndrome, sleep apnea).
* Current use of sleep-tracking technology (e.g., wrist-worn trackers, rings, smartphone apps) that could influence sleep behavior or perception.

Women currently undergoing perimenopause or experiencing vasomotor symptoms (e.g., night sweats).

* Use of hormone therapy (estrogen, progesterone, phytoestrogens) within the last 3 months.
* Diagnosed psychiatric disorders including major depressive disorder with acute symptoms, bipolar disorder, generalized anxiety disorder with active symptoms, and PTSD with frequent nightmares.
* Diagnosed neurodegenerative or chronic pain disorders, including Parkinson's disease, Alzheimer's disease, or uncontrolled fibromyalgia.
* Regular prescribed stimulant use (e.g., amphetamines such as Adderall/Vyvanse; methylphenidate such as Ritalin/Concerta; modafinil/armodafinil).
* Current use of CNS-activating antidepressants (bupropion, fluoxetine, venlafaxine, sertraline).
* Current or recent use of cannabis or THC-containing products (recreational or medicinal marijuana, CBD with measurable THC, synthetic cannabinoids) within the past 30 days.
* Employment in jobs disrupting nighttime sleep (e.g., night shift, rotating shift, excessive travel).
* Current use of prescription sleep aids.
* Introduction of any new sleep-related supplements, medications, herbal remedies, or melatonin products during the study.
* Use of any prescription or OTC products with sedative properties (e.g., melatonin, diphenhydramine, doxylamine, valerian, ZzzQuil, Advil PM) within 4 weeks prior to enrollment or habitual use ≥3 times per week prior to enrollment unless investigator-approved.
* Allergy or sensitivity to any study product ingredients.
* Pregnant, breastfeeding, or trying to conceive during the study period.
* History of substance abuse.
* Heavy alcohol use (≥8 drinks/week for women or ≥15 drinks/week for men).
* Participation in another research study now or within the next 7 weeks.
* Any condition or behavior that, in the investigator's judgment, may interfere with study participation or data integrity.

Ages: 22 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Evening relaxation, sleep quality, and morning vitality | Days 1, 3, 7, 14, 30
  Assessed by subjective questionnaire

OTHER OUTCOMES:
Sleep quality | Days 7, 14, and 30
  Assessed by subjective questionnaire
Daytime Sleepiness | Days 1, 7, 14, and 30
  Assessed by subjective questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philip Sapp, PhD, MS, Principal Investigator — Athletic Greens - AG1
Locations (1):
- Alethios (Virtual Study Platform), San Francisco, California, United States